CLINICAL TRIAL: NCT00875212
Title: Effect of a Dentifrice Containing Calcium Glycerophosphate and Fluoride on the pH of Dental Biofilm in Vivo
Brief Title: Effect of Calcium Glycerophosphate (CaGP) - Fluoride Dentifrice on Dental Biofilm pH
Acronym: CAGP-F
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: CAPES, Coordination for the Improvement of Higher Education Personnel
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UFPB-CAPES_2005; CNPq?PIBIC?UFPB_2005
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2009-10-12 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Dental Caries
Keywords: Calcium glycerophosphate; Fluoride; Dentifrice; Biofilm; Dental caries
MeSH Terms: conditions — Dental Caries | interventions — Glycerophosphates; Fluorides; Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- dentifrice intervention (Experimental): 4 types of dentifrices were used in 4 different periods in a crossover study design.
  Interventions: Drug: calcium glycerophosphate; Drug: no active ingredient; Drug: fluoride; Drug: CAGP + fluoride

INTERVENTIONS:
Drug: calcium glycerophosphate — use of a dentifrice containing CaGP (0.13%) and no fluoride
  Other Names: CaGP
Drug: no active ingredient — dentifrice without calcium glycerophosphate and no fluoride
  Other Names: dentifrice only (placebo)
Drug: fluoride — use of a dentifrice containing fluoride (1500ppm) only
  Other Names: sodium fluoride
Drug: CAGP + fluoride — calcium glycerophosphate and fluoride dentifrice
  Other Names: Experimental dentifrice with CAGP + fluoride

SUMMARY:
The aim of this study was to investigate the buffering effect of a calcium glycerophosphate-fluoride (CaGP-F) dentifrice on in vivo dental biofilm after a cariogenic challenge and evaluate its probable 12-hour protective effect. Twelve young adults took part in this randomized, double blind, 14-day 4-phase crossover study. Between each phase, the volunteers had a 1-week wash-out period. Coded dentifrices were randomly assigned to the volunteers: A) no F and no CaGP; B) CaGP-only (0.13%); C) F-only (1500 ppm (ppm= parts per million of fluoride which is equivalent to mg/kg)); D) CaGP-F (0.13%, 1500 ppm, respectively). The pH measurements were taken from a single-site using a microelectrode, with salt bridge established by a 1M KCl (one molar potassium chloride) solution with a reference electrode. pH measurements were taken at 0 (baseline), 1, 7, 14 and 21 min (minutes) after a cariogenic challenge (10% w/v sucrose solution, %w/v = percent weight per volume). Four sets of measurements were carried out: (D0BS) before test dentifrice usage; (D01min) 1-min after test dentifrice usage; and (D712h) 7 days and (D1412h) 14 days using the test dentifrice, 12 hours (h)after brushing. Stephen curves and mean AUC (area under the curve) were obtained.

DETAILED DESCRIPTION:
Although the mechanisms of action of fluoride are reasonably understood, the mechanism of calcium phosphate and calcium glycerophosphate (CaGP) are still a matter of debate. It has been suggested that CaGP increases the phosphorus content in the biofilm and, as a result, the buffering capacity of the biofilm is intensified. The pH levels of the biofilm are maintained above the 5.0-5.5 range. This is above the critical range for enamel demineralization.

ELIGIBILITY:
Inclusion Criteria:

* to live in a non-fluoridated area
* to have at least 20 natural teeth
* signed a consent form agreeing to carefully follow the research instructions

Exclusion Criteria:

* presence of active caries lesions
* periodontal disease
* use of antibiotics/medication.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio C Sampaio, PhD, Principal Investigator — Federal University of Paraiba; Thiago S Carvalho, Master, Study Chair — Federal University of Paraiba
Locations (1):
- Health Science Centre at the Federal University of Paraiba, João Pessoa, Paraíba, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were dental students of the University. The recruitment locations were dental clinics of the faculty and laboratory facilities.
  The dates of recruitment included 2-3 months before starting the research in January 2006; and lasted for 2 months afterwards
Pre-assignment Details: As a pre-assignment procedure, all volunteers signed an informed consent. The the volunteers received a dental hygiene kit containing a toothbrush and a fluoride-free and calcium-free dentifrice as part of the 1-week wash-out period prior to group assignment.
Groups:
- Toothbrushing: The study was based on the use of dentifrices for daily oral hygiene in a crossover design. The volunteers were asked to use the placebo and test dentifrices for one week. During the study, the volunteers were instructed to brush their teeth normally until 3 days before the measurements. During these 3 days, they were instructed to brush only the occlusal surfaces of their teeth until 12 hours before the pH measurements, when they should stop brushing altogether for dental plaque pH evaluation.
Period: Placebo Dentifrice
Arm/Group | Toothbrushing
Started | 12
Completed | 12 (all participants completed this group)
Not Completed | 0
Period: CaGP Only Dentifrice
Arm/Group | Toothbrushing
Started | 12
Completed | 12
Not Completed | 0
Period: Fluoride Only Dentifrice
Arm/Group | Toothbrushing
Started | 12
Completed | 12
Not Completed | 0
Period: CaGP and Fluoride Dentifrice
Arm/Group | Toothbrushing
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Toothbrushing
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  Brazil | 12

OUTCOME MEASURES:

1. Primary Outcome: Minimum pH
Description: The dental biofilm pH was measured in vivo with the microtouch method, using a palladium microelectrode + reference electrode. Data represents the mean values of the lowest pH observed each time after the use of sucrose.
Time Frame: at 1 minute (minimum fermenting pH) or at 7 minutes
Population: The number of subjects were determined by a pilot study carried out in 3 volunteers. The study has a crossover design. Thus the 4 groups of dentifrices tested included the same subjects in a different time-measurement avoiding the influence of individual variables in the analysis.
Measure: Mean (Standard Deviation); unit: pH
Groups:
- Control: intervention of using a dentifrice of no active ingredient. The volunteers were asked to use the placebo dentifrices for one week. Throughout the study, the volunteers were instructed to brush their teeth normally up until 3 days before the measurements. During these 3 days, they were instructed to brush only the occlusal surfaces of their teeth until 12 hours before the pH measurements, when they should stop brushing altogether for dental plaque pH evaluation.
- Calcium Glycerophosphate: intervention of using a dentifrice containing only calcium glycerophosphate (CaGP)
- Fluoride: intervention of using a dentifrice with 1,500 ppm of fluoride
- Calcium Glycerophosphate and Fluoride: intervention of using a dentifrice containing fluoride and calcium glycerophosphate
Arm/Group | Control | Calcium Glycerophosphate | Fluoride | Calcium Glycerophosphate and Fluoride
Number analyzed (Participants) | 12 | 12 | 12 | 12
pH | 5.40 (0.60) | 5.48 (0.65) | 5.25 (0.77) | 5.70 (0.43)
Statistical Analysis 1: Comparison: Control vs Calcium Glycerophosphate vs Fluoride vs Calcium Glycerophosphate and Fluoride; The study was based on the use of dentifrices for daily oral hygiene in a crossover design. The null hyphothesis was no difference between pH values of the groups. The statistical analysis was by repeated measurements ANOVA; Test type: Superiority or Other; p = 0.001, ANOVA; repeated measure anova; Median Difference (Final Values) = 5.5, Standard Deviation 0.25 — The median value of each parameter (pH baseline, minimal pH) was obtained and these values were compared between each group
Statistical Analysis 2: Comparison: Control vs Calcium Glycerophosphate vs Fluoride vs Calcium Glycerophosphate and Fluoride; The comparison was based on mean and median values of plaque pH in different moments of cariogenic challenge. The null hypothesis was that no diference between the groups wil be found. The test hypothesis was that the experimental dentifrice of CaGP-F would provide a better control of plaque pH after 14 days of use; Test type: Superiority or Other; p = 0.001, ANOVA; repeated-measurements ANOVA; Median Difference (Final Values) = 5.5, Standard Deviation 0.1

2. Primary Outcome: Minimum pH After 14 Days of Use of Dentifrice
Description: measurement of pH obtained as described before. However, this time the biofilm was exposed to the dentifrices for a longer period (14 days).
Time Frame: 14 days
Population: The initial part of the work as a pilot study.
Measure: Mean (Standard Deviation); unit: pH
Groups:
- Control: use of a placebo dentifrice (no fluoride and no CaGP). The volunteers were asked to use the placebo dentifrices for more one week. Throughout the study, the volunteers were instructed to brush their teeth normally up until 3 days before the measurements. During these 3 days, they were instructed to brush only the occlusal surfaces of their teeth until 12 hours before the pH measurements, when they should stop brushing altogether for dental plaque pH evaluation.
- Calcium Glycerophosphate: intervention of using a CaGP dentifrice
- Fluoride: intrvention of using a 1,500 ppm fluoridated dentifrice
- Calcium Glycerophosphate and Fluoride: intervention of using a CaGP+Fluoride dentifrice
Arm/Group | Control | Calcium Glycerophosphate | Fluoride | Calcium Glycerophosphate and Fluoride
Number analyzed (Participants) | 12 | 12 | 12 | 12
pH | 4.78 (0.67) | 5.24 (0.83) | 5.25 (0.71) | 5.44 (0.59)
Statistical Analysis 1: Comparison: Control vs Calcium Glycerophosphate vs Fluoride vs Calcium Glycerophosphate and Fluoride; The groups were compared by repeated measurements anova. There was no power calculation, but a pilot study to check the minimal number necessary of subjects in order to find a signifcant difference between interventions; Test type: Superiority or Other; p = 0.01, ANOVA; repeated measurements ANOVA; Mean Difference (Final Values) = 5.5, Standard Deviation 0.25 — The difference of pH values between groups was above 1.0 unit

ADVERSE EVENTS:
Arm/Group | Toothbrushing
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
pH measurements of dental biofilms were difficult after continuous use of dentifrice because of reduced biofilm mass in contrast to baseline measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes